CLINICAL TRIAL: NCT01585675
Title: Specimen Banking From Patients With Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 04-0688.cc; P50CA058187 (NIH)
Record Dates: First submitted 2012-04-17; First posted 2012-04-26 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Neoplasms
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, blood, urine, and sputum, breath
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnosis/treatment of lung cancer: Specimen Banking

SUMMARY:
The primary objective of the protocol is to develop a comprehensive specimen banking program from patients with lung cancer for future translation research, which will enable the investigators to detect lung cancer earlier, develop better therapies and explore screening and prevention strategies.

DETAILED DESCRIPTION:
The aims of the study are as follows: 1) to continue to unravel the complex biology of lung cancer 2) to identify early detection and prognostic markers to guide therapeutic decision 3) to define markers of response and/or resistance to drug therapy, and 4) to identify new therapeutic and prevention targets.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are undergoing further testing for the diagnosis or treatment of lung cancer.
2. Oral and written informed consent

Exclusion Criteria:

1. Any individual who does not give oral and written consent for participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are undergoing further testing for the diagnosis or treatment of lung cancer.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2005-11-03 (Actual); Primary Completion 2035-07-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
Development of a comprehensive specimen banking program from patients with lung cancer for future translational research. | 6 years
  No statistical analysis will be applied to the overall collection of samples. Rather, each project that utilized tissue bank resources will require an appropriate statistical plan to be submitted along with the initial tissue request.

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan VanBokhoven, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States